CLINICAL TRIAL: NCT06079931
Title: The Efficacy of Babaodan Capsules in Preventing Radiation Pneumonitis in Locally Advanced Non-Small Cell Lung Cancer Patients: A Phase II Clinical Trial
Brief Title: The Efficacy of Babaodan Capsules in Preventing Radiation Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZDWY.ZYZLK.004
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-08

CONDITIONS: Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis

STUDY DESIGN:
Intervention Model Description: Simon's optimal two-stage design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Babaodan combined with standard concurrent chemoradiotherapy treatment group (Experimental): 60-66Gy/30-33F radiotherapy, 2Gy/dose; During radiation therapy, concurrent chemotherapy including paclitaxel 45 mg/m2 and carboplatin (AUC 2) was administered once a week on the first day. From the start of radiation therapy to the completion of concurrent chemoradiotherapy (CCRT) for 2 months, the patient took 2 capsules of Babaodan orally every day, tid (1.8 g/day). Systemic corticosteroids can be used in patients with acute radiation pneumonia with G ≥ 2.
  Interventions: Drug: Babaodan Capsule

INTERVENTIONS:
Drug: Babaodan Capsule — The patient received 66-66Gy/30-33F radiation therapy. During radiation therapy, concurrent chemotherapy includes receiving 45mg/m2 paclitaxel and carboplatin (AUC 2) once a week; From the start of radiation therapy to 2 months after the completion of CCRT, the patient takes 2 capsules of Babaodan orally every day, tid (1.8 g/day), and systemic corticosteroids can be used for acute radiation pneumonia patients with G ≥ 2.
  Other Names: Babaodan

SUMMARY:
Radiation pneumonitis (RP) is a common complication of radiotherapy for thoracic tumors, and the incidence rate of grade 2 or above RP is 20% -40%; The use of antibiotics after secondary bacterial infection due to radiation pneumonia or the use of systemic glucocorticoids for radiation pneumonia itself have significant adverse effects on the survival of NSCLC patients. At present, FDA has not approved drugs to prevent the occurrence of radiation pneumonia. traditional Chinese patent Babaodan (BBD) capsule has the effect of controlling macrophages to produce proinflammatory cytokines, such as significantly inhibiting the release of IL-6. Through prospective research, this study evaluates the incidence of symptomatic pneumonia (G ≥ 2) in the treatment of locally advanced non-small cell lung cancer with BBD combined with concurrent radiotherapy and chemotherapy.

DETAILED DESCRIPTION:
Radiation induced lung injury (RILI) is a common complication of chest radiation therapy, which can be divided into two stages, including radiation pneumonia (RP) and pulmonary fibrosis (RPF), with different clinical manifestations and occurrence times. According to the research report, the incidence rate of grade 2 or above RP is 20% -40%, and most patients have different degrees of pulmonary fibrosis in the late stage. Although these two stages are interdependent, they can be clearly separated in terms of time: RP occurs within 6 months after treatment (usually within 12 weeks), while RPF occurs after more than 1 year of treatment. RILI is believed to be caused by reactive oxygen species produced during the treatment process, which can lead to DNA damage and subsequent inflammatory reactions. After irradiation of alveolar type II cells and endothelial cells, they release pro-inflammatory cytokines, promote the activation and chemotaxis of inflammatory cells, induce macrophages to release profibrotic factors, and stimulate fibroblast proliferation to promote fibrosis.

Babaodan (BBD) capsule has the effects of clearing heat and dampness, promoting blood circulation and detoxification, and treating jaundice and pain. Its characteristics are recognized as common symptoms of infectious diseases and inflammation in modern medicine. It is widely used in clinical practice to treat viral hepatitis, cholecystitis, vascular colitis, and urinary tract infections. Studies have found that BBD has a therapeutic effect on endotoxin-induced sepsis by inhibiting NLRP3 mediated activation of inflammasomes. It has also been reported that in the animal and clinical experiments of COVID-19, BBD controls macrophages to produce a large number of proinflammatory cytokines, such as significantly inhibiting the release of IL-6, thus realizing the protective effect of excessive immune response. In addition, in vivo and in vitro research results indicate that BBD can enhance the anti-tumor effect of cisplatin on non-small cell lung cancer (NSCLC).

We initiated this Phase II study to evaluate the efficacy of BBD in reducing the incidence of symptomatic RP in LANSCLC patients receiving CCRT treatment. In this study, BBD was delivered during and after CCRT, assuming that BBD can alleviate the potential harmful effects of CCRT and regulate the severity of pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* （1）18 to 70 years；（2）Histologically/cytologically confirmed NSCLC；（3）ECOG ≤2；（4）Weight loss ≤10%；（5） Inoperable AJCC stage IIIA, or IIIB disease；（6）Neutrophils ≥1.5×10^9/L and platelets ≥100×10^9/L；（7）Adequate liver and renal function.

Exclusion Criteria:

* （1）Malignant pleural effusion；（2）Active uncontrolled infection；（3）Significant cardiovascular disease；（4）History of other malignancies；（5）Forced expiratory volume in 1 second <40% of normal；（6）Previous history of cervical and chest radiation therapy.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of radiation pneumonia with G ≥ 2 | 14 months
  We used Simon's optimal two-stage design: the first stage requires the recruitment of at least 6 participants, of which at least 4 do not develop symptomatic radiation pneumonia. Once the goal is achieved, the second stage begins, and at least 21 more participants are recruited to achieve a total sample size of 27 patients. Overall, if at least 22 people do not experience symptomatic radiation pneumonia, the treatment plan will be considered successful. Increase the sample size by 10% to prevent falling off and insufficient statistics, so we plan to include 30 people.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yat sen University, Study Director — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dang J, Li G, Ma L, Diao R, Zang S, Han C, Zhang S, Yao L. Predictors of grade >/= 2 and grade >/= 3 radiation pneumonitis in patients with locally advanced non-small cell lung cancer treated with three-dimensional conformal radiotherapy. Acta Oncol. 2013 Aug;52(6):1175-80. doi: 10.3109/0284186X.2012.747696. Epub 2012 Dec 3. PMID 23198719
- [Background] Xu Y, Zheng X, Bai X, Li P, Ma H, Wang J, Hu X, Chen M. Simultaneous integrated boost intensity-modulated radiotherapy for locally advanced non-small cell lung cancer in Chinese population: A retrospective study. Oncotarget. 2017 Jul 25;8(30):49084-49092. doi: 10.18632/oncotarget.17094. PMID 28467775
- [Background] McDonald S, Rubin P, Phillips TL, Marks LB. Injury to the lung from cancer therapy: clinical syndromes, measurable endpoints, and potential scoring systems. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1187-203. doi: 10.1016/0360-3016(94)00429-O. PMID 7713782
- [Background] Hanania AN, Mainwaring W, Ghebre YT, Hanania NA, Ludwig M. Radiation-Induced Lung Injury: Assessment and Management. Chest. 2019 Jul;156(1):150-162. doi: 10.1016/j.chest.2019.03.033. Epub 2019 Apr 15. PMID 30998908
- [Background] Barthelemy-Brichant N, Bosquee L, Cataldo D, Corhay JL, Gustin M, Seidel L, Thiry A, Ghaye B, Nizet M, Albert A, Deneufbourg JM, Bartsch P, Nusgens B. Increased IL-6 and TGF-beta1 concentrations in bronchoalveolar lavage fluid associated with thoracic radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):758-67. doi: 10.1016/S0360-3016(03)01614-6. PMID 14967431
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Lurienne L, Cervesi J, Duhalde L, de Gunzburg J, Andremont A, Zalcman G, Buffet R, Bandinelli PA. NSCLC Immunotherapy Efficacy and Antibiotic Use: A Systematic Review and Meta-Analysis. J Thorac Oncol. 2020 Jul;15(7):1147-1159. doi: 10.1016/j.jtho.2020.03.002. Epub 2020 Mar 12. PMID 32173463
- [Background] Scott SC, Pennell NA. Early Use of Systemic Corticosteroids in Patients with Advanced NSCLC Treated with Nivolumab. J Thorac Oncol. 2018 Nov;13(11):1771-1775. doi: 10.1016/j.jtho.2018.06.004. Epub 2018 Jun 20. PMID 29935305
- [Background] Sha S, Dong J, Wang M, Chen Z, Gao P. Risk factors for radiation-induced lung injury in patients with advanced non-small cell lung cancer: implication for treatment strategies. World J Surg Oncol. 2021 Jul 16;19(1):214. doi: 10.1186/s12957-021-02321-3. PMID 34271911
- [Background] Xia C, Shi W, Zhang Y, Ding L, Gao L, Wang Q, Shao L, Dong L, Gao Y. Prevention and treatment of radiation-induced lung injury. Future Med Chem. 2020 Dec;12(23):2161-2173. doi: 10.4155/fmc-2019-0162. Epub 2020 Nov 23. PMID 33225740
- [Background] Li YF, Sheng HD, Qian J, Wang Y. The Chinese medicine babaodan suppresses LPS-induced sepsis by inhibiting NLRP3-mediated inflammasome activation. J Ethnopharmacol. 2022 Jun 28;292:115205. doi: 10.1016/j.jep.2022.115205. Epub 2022 Mar 17. PMID 35307576
- [Background] Qian J, Xu H, Lv D, Liu W, Chen E, Zhou Y, Wang Y, Ying K, Fan X. Babaodan controls excessive immune responses and may represent a cytokine-targeted agent suitable for COVID-19 treatment. Biomed Pharmacother. 2021 Jul;139:111586. doi: 10.1016/j.biopha.2021.111586. Epub 2021 Apr 8. PMID 33866132
- [Background] Wang Q, Liu Z, Du K, Liang M, Zhu X, Yu Z, Chen R, Qin L, Li Y, Zheng Y. Babaodan inhibits cell growth by inducing autophagy through the PI3K/AKT/mTOR pathway and enhances antitumor effects of cisplatin in NSCLC cells. Am J Transl Res. 2019 Aug 15;11(8):5272-5283. eCollection 2019. PMID 31497240